CLINICAL TRIAL: NCT06017037
Title: REward Processing And Citalopram Study
Acronym: REPAC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REPAC01
Record Dates: First submitted 2023-05-15; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-05

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citalopram (Experimental): Citalopram 20mg p.o. once daily for 7-9 days
  Interventions: Drug: Citalopram 20mg
- Placebo (Placebo Comparator): Lactose p.o. once daily for 7-9 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram 20mg — Citalopram 20mg tablets, encapsulated to aid blinding. To take per oral once daily for 7-9 days
  Arms: Citalopram
Drug: Placebo — Lactose monohydrate tablets encapsulated to aid blinding. To take per oral once daily for 7-9 days
  Arms: Placebo

SUMMARY:
The goal of this experimental medicine study is to examine the effect of increasing serotonin on reward processing in healthy volunteers. The main questions it aims to answer are:

1. Does a subacute increase in serotonin influence the activation regions during reward learning
2. Does a subacute increase in serotonin influence behavioural markers of reward valuation (effort task), responsiveness (taste task) and learning (learning task)

Participants will be:

given a 7-day course of the selective serotonin reuptake inhibitor, citalopram. undergo behavioural testing complete a reward learning task whilst undergoing fMRI

Researchers will compare results against a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Aged between 18 to 65 years
* Sufficient knowledge of English language to understand and complete study tasks

Exclusion Criteria:

* Current or past probable diagnosis of psychiatric illness, according to DSM-5 criteria, requiring intervention by a healthcare professional, including but not limited to psychosis, bipolar disorder, major depression, OCD, PTSD, substance abuse disorder or any eating disorder
* Current or past diagnosis of any significant personality disorder (e.g. borderline personality disorder) according to self-report
* Diagnosis of attention deficit hyperactive disorder or autistic spectrum disorder that impairs daily functioning, requires pharmacotherapy or in the opinion of the study medic would affect the scientific integrity of the study
* Current use of medication that might interact with the effects of citalopram or affect the scientific integrity of the study
* Previous suicide attempt or previous prolonged period (e.g. > 5 days) of thoughts to end life
* Known contraindication to citalopram including: past allergic reaction to citalopram or any other medicines, diagnosis of a cardiovascular condition, glaucoma, type 1 or type 2 diabetes, diagnosis of epilepsy, previous diagnosis of angle-closure glaucoma, or current use of any other medication whose use interacts with citalopram (according to BNF guidance) e.g. associated with prolonged QT-interval
* Any other current or past medical conditions which in the opinion of the study medic may interfere with the safety of the participant or the scientific integrity of the study including epilepsy/seizures, brain injury, hepatic or renal disease, diabetes, severe gastro-intestinal problems, Central Nervous System (CNS) tumours, neurological conditions
* First-degree relative with a diagnosis of schizophrenia-spectrum or other psychotic disorder, or bipolar disorder
* Severely underweight (BMI<17) or very obese (BMI>40) in a manner that renders them unsuitable for the study in the opinion of the study medic
* Heavy use of cigarettes (smoke > 20 cigarettes per day)
* Heavy use of caffeine (drink > 4 250ml cups/cans of coffee/energy drinks per day)
* Lactose intolerance (due to the study involving administration of a lactose placebo tablet)
* Known allergy to citric acid, sodium chloride, sucrose or quinine
* Pregnancy (as determined by urine pregnancy test taken during the Part 2 screening visit), breast feeding or plans to become pregnant
* past history of dependence on illicit substances or regular illicit substance use within previous three months
* Evidence of current or past harmful use of alcohol
* previous participation in a study involving the tasks used in this study or involving use of citalopram in the last year
* physical (including visual and auditory) or language impairment that would make complying with the study protocol challenging
* ongoing deficit in sense of smell or taste e.g. following Covid-19 infection
* Participant is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator
* Not suitable for MRI neuroimaging e.g. claustrophobia, difficulty remaining still for duration of scan
* Any MRI contraindications outlined in FMRIB 3 Tesla scanning safety form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Reward & aversive learning: behavioural correlates | Day 7-9 of treatment
  Optimal choice learning rate of conditioned stimuli to win and loss outcomes.
  During an instrumental reinforcement learning task participant will complete trials with a pair of symbols (the valence will either be loss or win, which is implicit).
  One symbol will be high chance of that outcome (either win or loss depending on the valence of the pair) and the other low chance of the outcome.
  In the win pair the optimal choice is the high chance symbol (i.e. to win), in the loss pair the optimal choice is the low chance option (i.e. avoid loss).
  In each allocation group the proportion of participants making an optimal choice will be calculated on a trial-by-trial basis. This provide the learning rate outcome.
Reward & aversive learning: neural correlates | Day 7-9 of treatment
  Activity of a network of brain regions associated with reward learning (during anticipation and outcome), in response to a positive & negative outcomes in reward learning task.
  This will be the difference in BOLD activation in certain brain regions (pertinent to reward processing) between allocation groups during the anticipation stage and the outcome stage of the instrumental learning task.

SECONDARY OUTCOMES:
Resting state | Day 7-9 of treatment
  Resting state fMRI activation
Subjective rating of primary reward | Day 0 and day 7-9 of treatment
  Subjective rating of four tastes (sweet, salt, sour & bitter) in terms of intensity, anticipation of pleasurableness and actual pleasurableness.
Reward & aversive learning: behavioural volatile reward learning task: total money won | day 7-9 of treatment
  Amount of money won/lost & total amount of money received.
Motivational reward task | day 7-9 of treatment
  Participants are asked to accept or decline hypothetical offers made of various combinations of reward and physical effort (grip strength). For a limited number of offers participants are asked to actually expend effort for offers too. The investigators will examine
  1. Proportion of offer acceptance for various levels of reward and effort
  2. proportion of accepted offers successfully obtained
Reward & aversive learning: behavioural volatile reward learning task: learning rate | day 7-9 of treatment
  Learning rate of optimal choices changes during the task. Proportion of participants in each allocation arm making an optimal choice on a trial-by-trial basis will provide the learning rate for each group.
  Provides sensitive measure of reward and aversive learning rates.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, PhD, Principal Investigator — University of Oxford
Locations (1):
- Neurosciences building, Department of Psychiatry, Warneford hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be anonymised and then processed for analysis. Anonymised data will be made available post-publication on Open Science Framework (OSF).
  defaced neural images will be shared via governed access through Zenodo with data sharing agreements in place